CLINICAL TRIAL: NCT07228884
Title: Improving Patient Comfort Without Sedation: The Impact of Verbal Suggestion on Anxiety and Pain During Colonoscopy
Brief Title: Verbal Suggestion to Reduce Pain and Anxiety During Unsedated Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasemin Keskin, Specialist in General Surgery, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-03/54
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Pain; Colonoscopy; Patient Comfort; Sedation-Free Procedure
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Suggestion Group (Experimental): Patients undergoing unsedated colonoscopy will receive positive verbal suggestion from the endoscopist throughout the procedure (e.g., "You are doing great," "Take a deep breath," "It will be over soon.")
  Interventions: Behavioral: Verbal Suggestion
- Control Group (No Intervention): Patients undergoing unsedated colonoscopy will receive standard communication without verbal suggestion during the procedure.

INTERVENTIONS:
Behavioral: Verbal Suggestion — During unsedated colonoscopy, the endoscopist will use positive verbal suggestions aimed at reducing patients' anxiety and perceived pain. The phrases include encouraging and calming statements such as "You are doing well," "Take a deep breath," and "We're almost done." The communication is supportive, consistent, and non-directive throughout the procedure.
  Arms: Verbal Suggestion Group

SUMMARY:
Colonoscopy is an important diagnostic and screening procedure for colorectal diseases, but it can cause pain and anxiety, especially when performed without sedation. Verbal suggestion techniques - in which the physician provides calm, positive, and encouraging communication during the procedure - may help reduce these unpleasant experiences.

This randomized controlled study aims to evaluate the effect of verbal suggestion on pain and anxiety levels of patients undergoing unsedated colonoscopy. Sixty adult patients will be randomly assigned to either a verbal suggestion group or a control group. In the verbal suggestion group, the endoscopist will use positive and supportive phrases during the procedure (for example: "You are doing great," "Take a deep breath, we'll get through this easily"). The control group will undergo colonoscopy without any verbal intervention.

Pain will be assessed using a Visual Analog Scale (VAS) and anxiety will be measured with the Beck Anxiety Inventory (BAI) before and after the procedure. Heart rate will also be monitored as an objective indicator of anxiety.

The goal of this study is to determine whether verbal suggestion can improve patient comfort and tolerance during colonoscopy without sedation, potentially providing a low-cost and practical method to enhance patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years.
* Patients scheduled for elective, diagnostic, or screening colonoscopy without sedation.
* Ability to understand and provide written informed consent.
* Ability to communicate verbally with the endoscopist during the procedure.
* ASA (American Society of Anesthesiologists) physical status classification I-II.

Exclusion Criteria:

* Refusal or inability to provide informed consent.
* Known psychiatric or neurological disorders that could affect anxiety or pain perception.
* Use of anxiolytic, sedative, or analgesic drugs within 24 hours before the procedure.
* Colonoscopy performed under sedation or anesthesia.
* Severe cardiopulmonary comorbidities (ASA class ≥ III).
* Incomplete colonoscopy due to technical or anatomical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Pain score during colonoscopy | immediately after procedure
  Pain intensity will be measured using the Visual Analog Scale (VAS; 0-10, higher scores indicate worse pain). The score will be recorded immediately after the procedure.

SECONDARY OUTCOMES:
Heart rate change during the procedure | During colonoscopy
  Heart rate will be monitored continuously during colonoscopy. The maximum heart rate recorded during the procedure will be used as an objective physiologic measure.
Anxiety level before and after colonoscopy | within 30 minutes before and after procedure
  ty will be assessed using the Beck Anxiety Inventory (BAI; 0-63, higher scores indicate greater anxiety). Pre- and post-procedure scores will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara, Yenimahalle, Turkey (Türkiye)